CLINICAL TRIAL: NCT06667128
Title: Optimization of Heart Failure (HF) Medical Therapy After Transcatheter Valve Intervention (TVI) in Patients With Heart Failure With Reduced Ejection Fraction (HFrEF)
Acronym: OPTIMAV
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Ospedale San Raffaele (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Principal Investigator, Cosmo Godino, Doctor (Co-PI), IRCCS Ospedale San Raffaele
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22071997
Record Dates: First submitted 2024-10-25; First posted 2024-10-31 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Heart Failure; Valvulopathy; Aortic Stenosis; Aortic Regurgitation Disease; Mitral Regurgitation; Tricuspid Regurgitation; Brain Natriuretic Peptide; Mitraclip; TAVI(Transcatheter Aortic Valve Implantation)
Keywords: Heart Failure; Aortic Stenosis; Aortic Regurgitation; Mitral Regurgitation; Tricuspid Regurgitation; Mitraclip; Triclip; TAVI
MeSH Terms: conditions — Heart Failure; Heart Valve Diseases; Aortic Valve Stenosis; Mitral Valve Insufficiency; Tricuspid Valve Insufficiency; Aortic Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Care Group (No Intervention): Participants receive standard follow-up care with Guideline-Directed Medical Therapy (GDMT) adjustments as per the physician's usual practice.
- Rapid Up-Titration GDMT Group with Point-of-Care (PoC) Monitoring (Experimental): Patients will undergo rapid up-titration of GDMT. Their progress will be closely monitored using Point-of-Care (PoC) technology from Roche Diagnostics for NT-proBNP measurements.
  Interventions: Other: Rapid Uptitration of Guideline-Directed Medical Therapy; Diagnostic Test: Elecsys® NT-proBNP - Roche Diagnostics
- Rapid Up-Titration GDMT Group with Hospital Monitoring (Experimental): Patients will undergo rapid up-titration of GDMT. Their progress will be closely monitored using hospital-based blood tests (Roche Elecsys central laboratory platform).
  Interventions: Other: Rapid Up-Titration GDMT Group with Hospital Monitoring

INTERVENTIONS:
Other: Rapid Uptitration of Guideline-Directed Medical Therapy — Rapid up-titration of GDMT guided by protocol-specific guideline.
  Arms: Rapid Up-Titration GDMT Group with Point-of-Care (PoC) Monitoring
Diagnostic Test: Elecsys® NT-proBNP - Roche Diagnostics — An assay provided by Roche (Elecsys® NT-proBNP - Roche Diagnostics) will be used to assess NT-proBNP levels in the Rapid Up-Titration GDMT Group with Point-of-Care (PoC) Monitoring, with the purpose of evaluating any differences in marker dosage between the indicated method and the monitoring by the hospital laboratory analysis.
  Other Names: Point-of-Care (PoC) Monitoring
  Arms: Rapid Up-Titration GDMT Group with Point-of-Care (PoC) Monitoring
Other: Rapid Up-Titration GDMT Group with Hospital Monitoring — Rapid Up-Titration GDMT Group guided by protocol-specific guideline and hospital monitoring.
  Arms: Rapid Up-Titration GDMT Group with Hospital Monitoring

SUMMARY:
This trial is a single-center, open-label, randomized study designed to assess the impact of a rapid up-titration of Guideline-Directed Medical Therapy (GDMT) on heart failure with reduced ejection fraction (HFrEF) patients following transcatheter valve interventions. The study focuses on the efficacy of intensive treatment in decreasing NT-proBNP levels and improving patient outcomes, including survival rates and quality of life over a six-month period. Patients are closely monitored using both Point-of-Care technology and hospital-based assessments, with the goal of enhancing GDMT adjustments. This approach is compared to standard care to determine its potential benefits in the management of HFrEF post-valve intervention.

DETAILED DESCRIPTION:
Heart valve disease, with a current prevalence of 2.5% that rises with age, has been described as "the next cardiac epidemic", and is projected to double by 2040 and triple by 2060, paralleling population aging.

The period during and immediately after hospitalization for transcatheter valve intervention (TVI) in HFrEF patients (LVEF ≤ 40%) represents a "vulnerable phase" characterized by a high risk of death and re-hospitalization for acute HF. A study from the TVI registry demonstrated that, among 12.182 patients treated with TAVR in the United States, the rate of HF readmission at 1 year was 14.3% and the 1-year overall mortality was 23.7%.

Moreover, the CHOICE-MI registry demonstrated that the primary combined endpoint of all-cause mortality or HF hospitalization at 1 year occurred in 39.2% of the Transcatheter mitral valve implantation (TMVI) patients, and in 28% in those TMVI-ineligible who undergoing bailout-TEER.

Recently, the STRONG-HF trial demonstrated that rapid, intensive up-titration of guideline-directed therapy, coupled with close post-discharge follow-up, significantly enhances life quality and reduces 180-day mortality and heart failure readmission rates versus usual care.

Previous studies have additionally shown that a decrease in NT-proBNP levels during hospitalization for acute HF is associated with improved survival and reduced readmission rates. Patients whose NT-proBNP levels decrease by at least 30% tend to have a better prognosis compared to those with no significant change or an increase in levels. This suggests that a meaningful decrease in NT-proBNP levels can indicate successful response to HF treatment.

Consequently, guiding HF therapy based on NT-proBNP levels can potentially improve clinical outcomes. For instance, adjusting medications to achieve a target NT-proBNP level may result in better control of HF symptoms and a lower risk of hospital readmission and mortality. This approach emphasizes the role of NT-proBNP as not just a diagnostic and prognostic tool but also as a therapeutic target in HF management. Overall, the use of NT-proBNP monitoring to guide medical therapy in HF patients supports a more personalized treatment strategy, potentially leading to rapid and effective decongestion, optimized therapy, and improved patient outcomes.

Hence, the primary objective of this study is to assess the impact of rapid up-titration of Guideline-Directed Medical Therapy (GDMT) in patients with HFrEF undergoing transcatheter valvular intervention, supplemented by close follow-up visits and NT-proBNP measurements, using a hierarchical composite endpoint, which prioritize (1) all-cause mortality, (2) number of hospitalizations for heart failure, and (3) improvement in NT-proBNP, defined as a decrease of at least 30% from the baseline value.

ELIGIBILITY:
Inclusion Criteria:

* Hospital admission for severe symptomatic valve disease (aortic stenosis, mitral regurgitation, or tricuspid regurgitation) effectively treated with transcatheter valve intervention (TVI) during hospitalization.
* Chronic heart failure with reduced ejection fraction (HFrEF)
* At the time of randomization (1-2 days prior to discharge):

  1. NT-proBNP > 900 pg/mL.
  2. Systolic blood pressure ≥ 100 mmHg.
  3. Heart rate ≥ 60 bpm.
  4. Serum potassium ≤ 5.0 mEq/L (mmol/L).
* At the time of hospital admission treated with ≤ ½ of the of optimal dose of ACEi/ARB/ARNi, ≤ ½ of the of optimal dose of beta-blocker, and ≤ ½ of the of optimal dose of MRA, either with or without SGLT2ic.
* Residency in the Lombardy region.
* Written informed consent to participate in the study.

Exclusion Criteria:

* Age < 18 or > 85 years.
* Clearly documented intolerance to ACEi/ARB/ARNI, or beta-blockers, or MRA, or SGLT2i.
* Residual severe valve disease of the valve treated with TVI (i.e. severe aortic stenosis or severe paravalvular leak after TAVR, severe mitral stenosis or severe residual mitral regurgitation after mitral valve intervention, or severe tricuspid stenosis or severe residual tricuspid regurgitation after tricuspid valve intervention).
* Presence at the time of randomization (1-2 days prior to discharge) of any severe valve disease.
* Hemodynamically significant obstructive lesion of the left ventricular outflow tract.
* Significant pulmonary disease contributing substantially to the patients' dyspnea such as FEV1< 1 liter or need for chronic systemic or non-systemic steroid therapy, or any kind of primary right HF such as primary pulmonary hypertension or recurrent pulmonary embolism.
* Myocardial infarction, unstable angina or cardiac surgery within 3 months, or cardiac resynchronization therapy device implantation within 3 months, or percutaneous transluminal coronary intervention, within 1 month prior to screening.
* Uncorrected thyroid disease, active myocarditis, or known amyloid or hypertrophic obstructive cardiomyopathy.
* History of heart transplant or on a transplant list or using or planned to be implanted with a ventricular assist device.
* Sustained ventricular arrhythmia with syncopal episodes within the 3 months prior to screening that is untreated.
* Active infection at any time during hospitalization requiring intravenous antibiotics.
* Stroke or TIA within 3 months prior to screening.
* Primary liver disease considered to be life threatening.
* Renal disease or eGFR < 30 mL/min/1.73m2 (as estimated by the simplified MDRD formula) at screening or history of dialysis.
* Psychiatric or neurological disorder, cirrhosis, or active malignancy leading to a life expectancy <12 months.
* Prior (defined as less than 30 days from screening) or current enrollment in a CHF trial or participation in an investigational drug or device study within the 30 days prior to screening.
* Discharge to a rehabilitation of long-term care facility.
* Inability to comply with all study requirements, due to major co-morbidities, social or financial issues, or a history of noncompliance with medical regimens, that might compromise the patient's ability to understand and/or comply with the protocol instructions or follow-up procedures
* Pregnant or nursing (lactating) women.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Composite Hierarchical Outcome for Mortality, Heart Failure Hospitalization, and NT-proBNP Response | From enrollment to the end of treatment (up to 6 months).
  Hierarchical composite endpoint composed of (1) all-cause death, (2) number of HF hospitalization, (3) improvement of NT-proBNP (with an improvement defined as a decrease of at least 30% from baseline).

SECONDARY OUTCOMES:
Incidence of cardiovascular death | From enrollment to the end of treatment (up to 6 months).
  The incidence of death attributable to cardiovascular causes, including sudden cardiac death, myocardial infarction, or worsening heart failure.
Rate of Heart Failure Readmission | From enrollment to the end of treatment (up to 6 months).
  The rate of hospital readmission due to worsening heart failure symptoms, requiring inpatient care following discharge from the initial intervention.
Composite endpoint of Heart Failure Readmission or All-Cause Death | From enrollment to the end of treatment (up to 6 months).
  A composite endpoint measuring the incidence of either heart failure-related hospital readmission or death from any cause.
Change in Quality of Life according to the European Heart Failure Self-care Behaviour Scale | From enrollment to the end of treatment (up to 6 months).
  Assessment of patient-reported quality of life changes using the European Heart Failure Self-care Behaviour Scale (EHFScBS), a 9-items scale where higher score means worse self care (possible range 9 - 45).
Change in Quality of Life according to the Kansas City Cardiomyopathy Questionnaire | From enrollment to the end of treatment (up to 6 months).
  Assessment of patient-reported quality of life changes using the Kansas City Cardiomyopathy Questionnaire (KCCQ), a validated health status measure for patients with heart failure. It contains four subdomains: Physical Limitation, Symptom Frequency, Quality of Life, and Social Limitations. Each subdomain provides an individual score from 0 to 100, with 0 denoting the worst and 100 the best possible health status.
Changes in NT-proBNP Levels | From enrollment to the end of treatment (up to 6 months).
  Evaluation of the reduction in NT-proBNP levels from baseline to study completion as a biomarker of heart failure status improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Maisano, Head of Cardiac Surgery, Principal Investigator — IRCCS Ospedale San Raffaele
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vahanian A, Beyersdorf F, Praz F, Milojevic M, Baldus S, Bauersachs J, Capodanno D, Conradi L, De Bonis M, De Paulis R, Delgado V, Freemantle N, Gilard M, Haugaa KH, Jeppsson A, Juni P, Pierard L, Prendergast BD, Sadaba JR, Tribouilloy C, Wojakowski W; ESC/EACTS Scientific Document Group. 2021 ESC/EACTS Guidelines for the management of valvular heart disease. Eur Heart J. 2022 Feb 12;43(7):561-632. doi: 10.1093/eurheartj/ehab395. No abstract available. PMID 34453165
- [Background] McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Skibelund AK; ESC Scientific Document Group. 2023 Focused Update of the 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure. Eur Heart J. 2023 Oct 1;44(37):3627-3639. doi: 10.1093/eurheartj/ehad195. No abstract available. PMID 37622666
- [Background] Bettencourt P, Azevedo A, Pimenta J, Frioes F, Ferreira S, Ferreira A. N-terminal-pro-brain natriuretic peptide predicts outcome after hospital discharge in heart failure patients. Circulation. 2004 Oct 12;110(15):2168-74. doi: 10.1161/01.CIR.0000144310.04433.BE. Epub 2004 Sep 27. PMID 15451800
- [Background] Adamo M, Pagnesi M, Mebazaa A, Davison B, Edwards C, Tomasoni D, Arrigo M, Barros M, Biegus J, Celutkiene J, Cerlinskaite-Bajore K, Chioncel O, Cohen-Solal A, Damasceno A, Diaz R, Filippatos G, Gayat E, Kimmoun A, Lam CSP, Novosadova M, Pang PS, Ponikowski P, Saidu H, Sliwa K, Takagi K, Ter Maaten JM, Voors A, Cotter G, Metra M. NT-proBNP and high intensity care for acute heart failure: the STRONG-HF trial. Eur Heart J. 2023 Aug 14;44(31):2947-2962. doi: 10.1093/eurheartj/ehad335. PMID 37217188
- [Background] Mebazaa A, Davison B, Chioncel O, Cohen-Solal A, Diaz R, Filippatos G, Metra M, Ponikowski P, Sliwa K, Voors AA, Edwards C, Novosadova M, Takagi K, Damasceno A, Saidu H, Gayat E, Pang PS, Celutkiene J, Cotter G. Safety, tolerability and efficacy of up-titration of guideline-directed medical therapies for acute heart failure (STRONG-HF): a multinational, open-label, randomised, trial. Lancet. 2022 Dec 3;400(10367):1938-1952. doi: 10.1016/S0140-6736(22)02076-1. Epub 2022 Nov 7. PMID 36356631
- [Background] Ben Ali W, Ludwig S, Duncan A, Weimann J, Nickenig G, Tanaka T, Coisne A, Vincentelli A, Makkar R, Webb JG, Akodad M, Muller DWM, Praz F, Wild MG, Hausleiter J, Goel SS, von Ballmoos MW, Denti P, Chehab O, Redwood S, Dahle G, Baldus S, Adam M, Ruge H, Lange R, Kaneko T, Leroux L, Dumonteil N, Tchetche D, Treede H, Flagiello M, Obadia JF, Walther T, Taramasso M, Sondergaard L, Bleiziffer S, Rudolph TK, Fam N, Kempfert J, Granada JF, Tang GHL, von Bardeleben RS, Conradi L, Modine T; CHOICE-MI Investigators. Characteristics and outcomes of patients screened for transcatheter mitral valve implantation: 1-year results from the CHOICE-MI registry. Eur J Heart Fail. 2022 May;24(5):887-898. doi: 10.1002/ejhf.2492. Epub 2022 Apr 17. PMID 35338542
- [Background] Holmes DR Jr, Brennan JM, Rumsfeld JS, Dai D, O'Brien SM, Vemulapalli S, Edwards FH, Carroll J, Shahian D, Grover F, Tuzcu EM, Peterson ED, Brindis RG, Mack MJ; STS/ACC TVT Registry. Clinical outcomes at 1 year following transcatheter aortic valve replacement. JAMA. 2015 Mar 10;313(10):1019-28. doi: 10.1001/jama.2015.1474. PMID 25756438